CLINICAL TRIAL: NCT03194282
Title: Effects of the Insole on Balance Capacity in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: N201705003
Record Dates: First submitted 2017-05-31; First posted 2017-06-21 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2018-05

CONDITIONS: Stroke, Cardiovascular
Keywords: stroke; balance; insole
MeSH Terms: conditions — Myocardial Infarction; Stroke | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic stroke patient with insole (Experimental): Poor balance capacity is one of clinical symptoms of stroke patient.Poor balance, or postural stability, is significant predictors the risk of fall.
  Interventions: Other: insole
- chronic stroke patient without insole (Sham Comparator): Poor balance capacity is one of clinical symptoms of stroke patient.Poor balance, or postural stability, is significant predictors the risk of fall.
  Interventions: Other: insole

INTERVENTIONS:
Other: insole — The subjects are randomly assigned to assess balance capacity either with or without insole.

SUMMARY:
Poor balance capacity is one of clinical symptoms of stroke patient. The reason of loss balance capacity is motor impairment, as well as a diminished capacity to voluntarily shift body weight or to with stand external pertubations. Postural movement patterns include three discrete control strategies: hip, knee, and ankle strategy. The ankle rocker is an important factor to maintain balance during standing and the ankle strategy restores the center of mass (CoM) to a position of stability through body movement. As a result, effective control of foot motion and ankle stability may decrease postural sway and the risk of fall in chronic stroke.The purpose of this study is to investigate the effects of the insole on balance capacity in chronic stroke.

DETAILED DESCRIPTION:
An important determinant of activities of daily living performance is standing balance. Therefore, poor balance, or postural stability, is significant predictors the risk of fall. After a fall, the patient can experience psychological, physical, social, economic, and sometimes fatal effects. The injuries can reduce the patient's mobility as well as independence and influence quality of life.Patients with chronic stroke wearing functional insoles and sham insoles to challenge balance tests.

ELIGIBILITY:
Inclusion Criteria:

* A history of unilateral chronic stroke occurrence over 6 months prior to the study
* Ability to understand verbal instructions.
* Ability to walk 5 meters independently without the need of ankle-foot orthosis.

Exclusion Criteria:

- A diagnosis of other neurological or musculoskeletal disorders that could affect postural balance.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Berg balance scale from pre to post-intervention. | up to 30 minutes.
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks.
Change in Functional Reach Test(FRT) from pre to post-intervention. | up to 10 minutes.
  The Functional Reach Test (FRT) is a quick screen for determining risk for falls.
Change in Timed Up and Go (TUG) Test from pre to post-intervention. | up to 10 minutes.
  Timed Up and Go (TUG) Test was developed to assess mobility.

SECONDARY OUTCOMES:
Change in Center of pressure (CoP) from pre to post-intervention. | up to 30 minutes.
  The center of pressure (CoP) measures derived from the foot pressure mat and force plate of Biodex Balance system.

CONTACTS AND LOCATIONS:
Overall Officials: YENTING LIU, Master, Study Chair — Wang Fang Hospital, Taipei Medical University
Locations (1):
- Wang Fang hospital, Taipei, Taipei City, Taiwan

REFERENCES:
- [Background] Christovao TC, Neto HP, Grecco LA, Ferreira LA, Franco de Moura RC, Eliege de Souza M, Franco de Oliveira LV, Oliveira CS. Effect of different insoles on postural balance: a systematic review. J Phys Ther Sci. 2013 Oct;25(10):1353-6. doi: 10.1589/jpts.25.1353. Epub 2013 Nov 20. PMID 24259792
- [Background] Chen TH, Chou LW, Tsai MW, Lo MJ, Kao MJ. Effectiveness of a heel cup with an arch support insole on the standing balance of the elderly. Clin Interv Aging. 2014 Feb 20;9:351-6. doi: 10.2147/CIA.S56268. eCollection 2014. PMID 24600215
- [Background] Rougier PR, Genthon N. Dynamical assessment of weight-bearing asymmetry during upright quiet stance in humans. Gait Posture. 2009 Apr;29(3):437-43. doi: 10.1016/j.gaitpost.2008.11.001. Epub 2008 Dec 12. PMID 19070493
- [Derived] Liu YT, Tsai HT, Hsu CY, Lin YN. Effects of orthopedic insoles on postural balance in patients with chronic stroke: A randomized crossover study. Gait Posture. 2021 Jun;87:75-80. doi: 10.1016/j.gaitpost.2021.04.014. Epub 2021 Apr 20. PMID 33894465